CLINICAL TRIAL: NCT01495403
Title: A Pilot Study of Hydroxychloroquine for the Treatment of Muscle Cramps in Patients With Cirrhosis
Brief Title: Treatment of Muscle Cramps in Patients With Liver Cirrhosis
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Patrick Kamath, PI, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 11-002743
Record Dates: First submitted 2011-12-16; First posted 2011-12-20 (Estimated); Last update posted 2023-05-03 (Actual); Status verified 2023-05

CONDITIONS: Liver Cirrhosis; Muscle Cramps
Keywords: liver cirrhosis; muscle cramps
MeSH Terms: conditions — Liver Cirrhosis; Muscle Cramp | interventions — Hydroxychloroquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- hydroxychloroquine (Experimental)
  Interventions: Drug: Hydroxychloroquine

INTERVENTIONS:
Drug: Hydroxychloroquine — daily dosing
  Other Names: Plaquenil

SUMMARY:
This is a pilot study to see if hydroxychloroquine (HCQ) if safe and effective to use with patients having cramps due to their cirrhotic liver disease.

DETAILED DESCRIPTION:
This project is proposed as a pilot study to gather preliminary data for a full-scale randomized trial to assess the efficacy and safety of hydroxychloroquine (HCQ) in the treatment of muscle cramps in patients with cirrhosis.

ELIGIBILITY:
Inclusion Criteria:

* previous diagnosis of cirrhosis
* adult (>21 years)
* able to complete a written questionnaire in English
* stable and ambulatory
* MELD score < 25, Platelet count >25,000

Exclusion Criteria:

* people allergic to hydroxychloroquine, 4-aminoquinolone derivatives or any component of the formulation
* previous diagnosis of retinal or visual field changes attributable to 4-aminoquinolone
* previous diagnosis of porphyria
* previous diagnosis of psoriasis
* fulminant hepatic failure
* pregnant women

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2011-12; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
frequency and severity of muscle cramps in cirrhotic patients reporting the symptom, based on the modified muscle cramps questionnaire (mMCQ) | 1 month after completion of questionnaire
  Patients will be given the mMCQ and SF-12 to complete. These instruments will be scored according to established algorithms. Data analysis will include descriptive statistics (frequency, duration and severity of muscle cramps) and correlation between overall quality of life and the mMCQ summary score.

SECONDARY OUTCOMES:
safety and efficacy of HCQ for severe cramping using mMCQ, SF-12, and AE inventory. | 28 days after first dose
  The study intervention will include open label HCQ daily, which will be provided for the patients for two weeks. A designated coordinator will contact the patient 2 and 7 days of the study to ask of adverse events and fill out the AE inventory. At the end of the dosing, patients will be asked to return to the clinic for post-intervention assessment, which will include the mMCQ, SF-12, systemic AE inventory, CBC and EKG. Designated coordinator will contact patient again on day 28 of the study to ask mMCQ, SF-12, AE inventory.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Kamath, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States